CLINICAL TRIAL: NCT00054600
Title: A Study of Extracorporeal Photopheresis With UVADEX in the Setting of a Standard Myeloablative Conditioning Regimen for the Prevention of Graft-versus-Host Disease in Patients Undergoing an Allogeneic Bone Marrow Transplant or Peripheral Blood Stem Cell Transplant
Brief Title: Safety and Efficacy Study of Photopheresis With UVADEX to Prevent Graft-versus-Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GvHD Prevention
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Graft-versus-Host Disease
Keywords: Extracorporeal Photopheresis; Graft-versus-Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Methoxsalen; Photopheresis

INTERVENTIONS:
Drug: Methoxsalen
Procedure: Extracorporeal Photopheresis

SUMMARY:
The purpose of this study is to determine whether Extracorporeal Photopheresis with UVADEX (ECP) prior to bone marrow or peripheral blood stem cell transplantation is effective in the prevention of Graft-versus-Host Disease (GvHD).

DETAILED DESCRIPTION:
Approximately 30% of HLA-identical related bone marrow graft recipients and up to 90% of patients receiving bone marrow from unrelated donors develop significant acute GvHD despite the use of prophylactic therapies such as cyclosporine and methotrexate. About half of these patients respond to initial treatment with steroids and require no further treatment. The remainder of these patients are either unresponsive to initial therapy or become steroid-resistant over time. The prognosis in these cases is poor and mortality for patients with steroid-resistant GvHD may be as high as 50%.

ECP is a technique in which peripheral white blood cells are exposed to a photoactivatable compound (UVADEX) administered extracorporeally and ultraviolet A light. After cells are reinfused into the patient, their function is altered, thereby activating mechanisms that allow for further regulation of specific lymphocyte populations. ECP has shown activity in several inflammatory and autoimmune diseases, including scleroderma, rheumatoid arthritis, transplantation rejection, acute and chronic GvHD.

In a previous single-center, open label, single-arm study of 56 patients receiving ECP treatment on two consecutive days and reduced-intensity bone-marrow conditioning prior to bone marrow transplantation from matched or partially matched human donors, the incidence of grade II-IV acute GvHD was less than 10%. This is in contrast to an expected incidence of approximately 40%.

The purpose of this study is to determine the role of ECP, administered pre-transplant, in preventing GvHD when used in conjunction with a standard myeloablative conditioning regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of a malignancy of the blood (e.g. leukemia) for which allogeneic bone marrow or peripheral blood stem cell transplantation is a treatment option.
* Patients who are candidates for a standard allogenic bone marrow transplant or PBSC transplant.
* Patients must have adequate renal, hepatic, pulmonary and cardiac function to enable the patient to tolerate shifts in the volumes of body fluids associated with extracorporeal photopheresis, as determined by the physician's clinical judgement.
* Patients must weigh at least 40 kg (88 lbs)

Exclusion Criteria:

* Patients who have received a prior bone marrow transplant or peripheral blood stem cell transplant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60
Dates: Start 2002-06; Study Completion 2004-06

CONTACTS AND LOCATIONS:
Locations (21):
- United States (6):
  - University of Florida, Gainesville, Florida
  - University of Chicago, Chicago, Illinois
  - Tufts New England Medical Center, Boston, Massachusetts
  - Kansas City Cancer Center, Kansas City, Missouri
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Texas Transplant, San Antonio, Texas
- Australia (5):
  - Royal Brisbane Hospital, Brisbane
  - Peter MacCallum Cancer Institute, East Melbourne
  - Alfred Hospital, Melbourne
  - Royal Melbourne Hospital, Parkville
  - St. Vincent's Hospital, Sydney
- Brazil (3):
  - Hospital Azevedo Carvalho, Jaú
  - National Cancer Institute, Rio de Janeiro
  - Hemocentro, São Paulo
- Ludwig-Maximiliano Universitaet Muenchen, München, Germany
- Italy (2):
  - Careggi Hospital, Florence
  - San Martino Hospital, Genova
- Instituto Portugues de Oncologia de Francisco Gentil, Lisbon, Portugal
- National Cancer Institute, Bratislava, Slovakia
- Ankara University Medical School, Ankara, Turkey (Türkiye)
- Hammersmith Hospital, London, United Kingdom

REFERENCES:
- [Background] Shlomchik WD, Couzens MS, Tang CB, McNiff J, Robert ME, Liu J, Shlomchik MJ, Emerson SG. Prevention of graft versus host disease by inactivation of host antigen-presenting cells. Science. 1999 Jul 16;285(5426):412-5. doi: 10.1126/science.285.5426.412. PMID 10411505